CLINICAL TRIAL: NCT04592900
Title: Virtual Reality Versus Biodex Balance Training In Adolescent Athletes With Chronic Ankle Instability.
Brief Title: Comparing VR and Balance Exercises In Rehabilitation of Adolescent Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Nehad Ahmed Youness Abo-zaid, Lecturer of physical therapy, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002877
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Sport Injury
Keywords: BalanceTraining,; Virtual Reality,; Ankle Instability.

STUDY DESIGN:
Intervention Model Description: G 1 (control) received traditional physical therapy program for 60 min. G 2(study) received traditional physical therapy program for 30 min. and virtual reality for 30 min. G 3 (study) received traditional physical therapy program for 30 min. and Biodex Balance Training all groups treated for four successive months.
Who Masked: Participant
Masking Description: Single (Outcomes Assessor) Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group 1 (control group) and Group 2 (virtual reality group), group 3 (Biodex Balance Training)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the control group (Experimental): the control group Group 1 the control group received selected physical therapy program which contain strengthening exercises for upper limb and lower limb muscles, stretching exercises for elbow extensors, hand supinator, wrist extensors, knee extensors and ankle dorsiflexors, balancing exercises, coordination exercises and balance training exercises and gait training in open environment.
  Interventions: Other: balance exercising
- the virtual reality group (Experimental): Group 2 the study group received the same physical therapy program 30 min. plus virtual reality for 30 min
  Interventions: Other: balance exercising
- the Biodex Balance Training group (Experimental): Group 3 the study group received the same physical therapy program 30 min. plus virtual reality for 30 min
  Interventions: Other: balance exercising

INTERVENTIONS:
Other: balance exercising — selected physical therapy program strengthening the muscles of upper and lower limbs, balancing exercise, gait training in open environment,stretching for elbow flexors and forearms pronators,lower limb hip flexors and knee extensor and ankle dorsiflexors

SUMMARY:
Ankle sprains are common injuries in active young people. Most of these injuries recovery quickly on their own, do not require imaging, and do better with early motion and rehabilitation. High ankle sprains and fractures are much less common but more serious. They may require imaging and more treatment.

DETAILED DESCRIPTION:
Phases of rehabilitation for ankle sprain Phase I treatment involves resting and protecting the ankle to permit healing, to prevent further injury, and to control pain and swelling.

Phase II treatment begins once pain and swelling have subsided to the point where the athlete can comfortably bear weight and walk from place to place.

Virtual reality (VR) is a simulated experience that can be similar to or completely different from the real world. Applications of virtual reality can include entertainment (i.e. video games) and educational purposes (i.e. medical or military training). Other, distinct types of VR style technology include augmented reality and mixed reality.

Biodex Balance Training is one of the main tool that used to assess dynamic balance and dynamic limits of stability also it can used as training tool to improve the participant balance training

ELIGIBILITY:
Inclusion Criteria:

1. Children will have sustained lateral ankle sprain (grade II).
2. Their age was ranging from 13-16 years
3. All children with stable medical and psychological status.
4. They will able to follow the verbal commands or instructions during testing.

Exclusion Criteria:

1. Children with ankle or foot deformity
2. Unstable medical and psychological status.
3. Children not able to follow the verbal commands or instructions during testing
4. Children with any disorder affecting balance.

Ages: 13 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — 90 boys were recruited and assesseted for eligability then randomly divided into 3 groups each one included 30 boy
Enrollment: 90 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
dynamic balance test | antro-posterior stability index at day 0
  antro-posterior stability index
dynamic balance test | antro-posterior stability index at day 90
  antro-posterior stability index
dynamic balance test | medio-lateral stability index at day 0
  medio-lateral stability index
dynamic balance test | medio-lateral stability index at day 90
  medio-lateral stability index
dynamic balance test | overall stability index at day 0
  overall stability index
dynamic balance test | overall stability index at day 90
  overall stability index

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A Abo-zaid, Principal Investigator — South Valley University, Faculty of Physical Therapy
Locations (1):
- Nehad Ahmed Youness, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pommering TL, Kluchurosky L, Hall SL. Ankle and foot injuries in pediatric and adult athletes. Prim Care. 2005 Mar;32(1):133-61. doi: 10.1016/j.pop.2004.11.003. PMID 15831316
- [Background] Waterman BR, Owens BD, Davey S, Zacchilli MA, Belmont PJ Jr. The epidemiology of ankle sprains in the United States. J Bone Joint Surg Am. 2010 Oct 6;92(13):2279-84. doi: 10.2106/JBJS.I.01537. PMID 20926721
- [Background] Hootman JM, Dick R, Agel J. Epidemiology of collegiate injuries for 15 sports: summary and recommendations for injury prevention initiatives. J Athl Train. 2007 Apr-Jun;42(2):311-9. PMID 17710181
- [Background] Williams MA, Soiza RL, Jenkinson AM, Stewart A. EXercising with Computers in Later Life (EXCELL) - pilot and feasibility study of the acceptability of the Nintendo(R) WiiFit in community-dwelling fallers. BMC Res Notes. 2010 Sep 13;3:238. doi: 10.1186/1756-0500-3-238. PMID 20831836
- [Background] Arifin N, Abu Osman NA, Wan Abas WA. Intrarater test-retest reliability of static and dynamic stability indexes measurement using the Biodex Stability System during unilateral stance. J Appl Biomech. 2014 Apr;30(2):300-4. doi: 10.1123/jab.2013-0130. Epub 2013 Jul 20. PMID 23878204

DOCUMENTS (1):
  • Study Protocol (2020-10-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT04592900/Prot_000.pdf